CLINICAL TRIAL: NCT04852731
Title: Dynamic Evaluation of Myocardial Fibrosis and Structural Determinants of Ventricular Arrhythmia in Mitral Valve Prolapse (STAMP-2 : STretch and Myocardial Characterization in Arrythmogenic Mitral Valve Prolapse-2)
Brief Title: STretch and Myocardial Characterization in Arrythmogenic Mitral Valve Prolapse-2
Acronym: STAMP-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Jean-Marc SELLAL, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02680-39
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Mitral Valve Prolapse
MeSH Terms: conditions — Mitral Valve Prolapse | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (a) : patients without mitral regurgitation without ventricular extrasystole (≤10/hour) (Experimental): These patients will undergo at the inclusion and 36 months after the inclusion :
  * According to recommendations : echocardiography, 24-hour external loop recording and exercise ECG,
  * And specifically for research purposes : injected cardiac MRI and a blood collection.
  Interventions: Procedure: Cardiac MRI; Other: Blood collection
- Group A (b) : patients without mitral regurgitation with ventricular extrasystole (>10/hour) (Experimental): These patients will undergo at the inclusion and 36 months after the inclusion :
  * According to recommendations : echocardiography, 24-hour external loop recording, exercise ECG, injected cardiac MRI,
  * And specifically for research purposes : prolongation of the MRI examination (4D flow sequence) and a blood collection.
  Interventions: Other: Blood collection; Procedure: Prolongation of the MRI examination
- Group B : patients with Mitral valve prolapse with trivial mitral regurgitation (Experimental): These patients will undergo at the inclusion and 36 months after the inclusion :
  * According to recommendations : echocardiography, 24-hour external loop recording, exercise ECG, injected cardiac MRI,
  * And specifically for research purposes : prolongation of the MRI examination (4D flow sequence) and a blood collection.
  Interventions: Other: Blood collection; Procedure: Prolongation of the MRI examination
- Group C : patients with Mitral valve prolapse with moderate or mild mitral regurgitation (Experimental): These patients will undergo at the inclusion and 36 months after the inclusion :
  * According to recommendations : echocardiography, 24-hour external loop recording, exercise ECG, injected cardiac MRI,
  * And specifically for research purposes : prolongation of the MRI examination (4D flow sequence) and a blood collection.
  Interventions: Other: Blood collection; Procedure: Prolongation of the MRI examination
- Group D : patients with asymptomatic Mitral valve prolapse with severe mitral regurgitation (Experimental): These patients will undergo at the inclusion and 36 months after the inclusion :
  * According to recommendations : echocardiography, 24-hour external loop recording, exercise ECG, injected cardiac MRI,
  * And specifically for research purposes : prolongation of the MRI examination (4D flow sequence) and a blood collection.
  Interventions: Other: Blood collection; Procedure: Prolongation of the MRI examination

INTERVENTIONS:
Procedure: Cardiac MRI — Injected cardiac MRI
  Arms: Group A (a) : patients without mitral regurgitation without ventricular extrasystole (≤10/hour)
Other: Blood collection — Blood collection (including genetics at the inclusion visit)
Procedure: Prolongation of the MRI examination — Prolongation of the MRI examination (4D flow sequence ; about 10 min)
  Arms: Group A (b) : patients without mitral regurgitation with ventricular extrasystole (>10/hour); Group B : patients with Mitral valve prolapse with trivial mitral regurgitation; Group C : patients with Mitral valve prolapse with moderate or mild mitral regurgitation; Group D : patients with asymptomatic Mitral valve prolapse with severe mitral regurgitation

SUMMARY:
Mitral valve prolapse (MVP) is a frequent affection of the mitral valve with a prevalence of 2-3% in the general population. This valvular disease is generally considered as benign, but may at term evolve toward mitral valve regurgitation of various severity and/or arrhythmia.

Mitral valve prolapse is routinely diagnosed using transthoracic echocardiography. Subsequent examinations (24-hour external loop recording, exercise electrocardiogram, cardiac Magnetic Resonance Imaging) and a close follow-up can be proposed to the patient depending on its condition.

More recently, detection of myocardial fibrosis and a mitral ring disjunction among patients with MVP were associated with the occurrence of severe ventricular arrhythmia.

The investigators hypothesize that ventricular remodeling over time is mediated by the progression of mitral insufficiency severity from myocardial fibrosis secondary to MVP and possibly promoted by other mitral valve abnormalities. This remodeling, characterized by circulating biomarkers and imaging (MRI and echocardiography), could allow the identification of patients with a higher risk of severe ventricular arrhythmia.

The main objective of this study is to identify prognostic factors for unfavorable evolution (ventricular remodeling or a rhythm disorder event) at 3 years from initial assessments in MVP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old,
* Patient with mitral valve prolapse,
* Patient who has received full information about the organization of the research and has signed an informed consent,
* Patient affiliated to or beneficiary of a social security insurance,
* Patient who has completed a prior clinical examination adapted to the research and who does not show any contraindication to the planned examinations

Exclusion Criteria:

* Stage of the disease: Patients with MVP with severe mitral regurgitation with a surgical indication as defined by current recommendations will not be included in the study,
* Presence of severe rhythm disorders requiring the implantation of a defibrillator (cardiorespiratory arrest recovered, sudden death recovered, etc.),
* Performance of an injected MRI in the month preceding the MRI scheduled during visit n°1,
* Previously diagnosed cardiopathy that may be responsible for myocardial damage (ventricular remodeling, alteration of left ventricular systolic function, fibrosis, etc.) and that may disrupt the interpretation of results (infarction, amyloidosis, systemic scleroderma, significant aortic valvulopathy, etc.).
* Contraindication to MRI examination, particularly in the presence of an implantable pacemaker or defibrillator, implanted pump, cochlear implants, neurosurgical clips, intraorbital or encephalic metallic foreign bodies,
* Claustrophobia or morphotype that does not allow MRI to be performed,
* Motor or mental disability,
* Renal impairment that does not allow the injection of Gadolinium-based contrast media (DOTAREM® or equivalent in the study). If there is any doubt as to the patient's renal function, a plasma creatinine determination will be performed for MRI to ensure the absence of renal failure,
* Hypersensitivity to gadoteric acid, meglumine, or any gadolinium-containing drug.
* Women of childbearing age who do not have effective contraception,
* Persons referred to in Articles L. 1121-5 to L1121-8 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Presence of ventricular remodelling | 3 years
  Variation of at least 10% of the telestolic volume observed at 3 years on cardiac MRI compared to the initial cardiac MRI
Presence of ventricular arrythmia (fibrillation or tachycardia, extrasystoles) | 3 years
  Occurrence of any ventricular arrythmia on external loop recording or exercise ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy University Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No